CLINICAL TRIAL: NCT06036823
Title: 5 Versus 10 Units of Insulin in Hyperkalemia Management: Multi-center, Prospective, Double-blind, Non-inferiority, Randomized Control Trial.
Brief Title: 5 Versus 10 Units of Insulin in Hyperkalemia Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Collaborators: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, Adnan Al-Ajmi, Doctor, Oman Medical Speciality Board
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MREC #2779
Record Dates: First submitted 2023-08-10; First posted 2023-09-14 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Hyperkalemia; Potassium Imbalance; Electrolyte Imbalance; Electrolyte Disturbance
Keywords: insulin; hyperkalemia; hypoglycmiea; anti-hyperkalemia; electrolytes abnormalities
MeSH Terms: conditions — Hyperkalemia; Insulin Resistance | interventions — Insulin; Albuterol

STUDY DESIGN:
Intervention Model Description: the study group will receive 5 units of intravenous insulin control group will receive 10 unites of IV insulin
Who Masked: Participant, Care Provider, Investigator
Masking Description: after consent. the care provider will take an envelope and give it to the nurse in charge of that patient without looking for the dose of insulin. as the same time will take the randomization code and stick it to the data collection sheet of that patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 5 units of intravenous R insulin (Active Comparator): Will receive:
  IV Insulin Regular 5 units with Dextrose 50 % 50 ml over 30 minutes. Salbutamol 10 mg Nebulization over 15 minutes.
  Interventions: Drug: Insulin regular; Drug: Dextrose 50; Drug: salbutamol
- 10 units of intravenous R insulin (Active Comparator): Will Receive:
  IV Insulin Regular 10 units with Dextrose 50 % 50 ml over 30 minutes. Salbutamol 10 mg nebulization over 15 minutes.
  Interventions: Drug: Insulin regular; Drug: Dextrose 50; Drug: salbutamol

INTERVENTIONS:
Drug: Insulin regular — Intravenous insulin
Drug: Dextrose 50 — to be given to both arms
Drug: salbutamol — to be given to all patients

SUMMARY:
The goal of this study is to compare 5 units of intravenous Regular insulin to 10 units of intravenous regular insulin in the management of hyperkalemia. We will measure the efficacy of these 2 doses of insulin in reducing hyperkalemia at 2 hours from administration using the main laboratory serum values.

DETAILED DESCRIPTION:
Introduction: Hyperkalaemia is a serum Potassium (K) level of more than 5.5 mEq/L. It is a common emergency medicine presentation and can be life-threatening. Because of the emergency in correcting hyperkalemia, different medications are used to reduce high potassium levels to normal as soon as possible. Salbutamol inhalers, Glucose solutions, and Insulin are the main medications for managing hyperkalemia. Insulin and Dextrose shift potassium ions into body cells by stimulating the sodium/potassium ATP pump. Its effect starts in less than fifteen minutes and can last up to sixty minutes. It usually reduces potassium up to 1.1 mEq/l. There are different recommendations for Insulin dose and rate of administration for patients with hyperkalemia.

Method: This will be a multi-center, prospective, double-blind, non-inferiority, randomized control trial. 336 hyperkalemia patients will be randomized to the intervention group 5 units of intravenous Regular insulin and 10 units of intravenous insulin groups with fifty ml of Dextrose Fifty percent. They will be enrolled once their potassium level is 5.5mEq/L or more. The attending physician and patient will be blinded about the dose of insulin that the patient received. Serum potassium will be measured at 0 and at 120 minutes from the start of the medications. Random blood glucose will be measured at 0, 60, and 120 minutes by Glucometer. The safety of our patients will be assessed by documentation of all adverse events, vital signs, and clinical assessment before and after drug administration. The study will end at 2 hours from insulin administration.

Aim: Our research idea aims to compare two recommended doses of Insulin (5 Units vs. 10 Units of Regular insulin given intravenously over thirty minutes) in the management of patients with hyperkalemia.

Primary objective: Mean reduction in serum potassium level using the main laboratory results at two hours from medication administration.

Secondary objectives: effect of initial (baseline) potassium level on the mean potassium reduction, and frequency of hypoglycemia between the 2 groups. Does the initial (baseline) blood glucose level will affect the function of insulin/dextrose in lowering potassium levels?

Patient Population: Adult patients (Aged 18 years and older) who present to the Emergency department at Sultan Qaboos University, Royal Hospital and Sohar hospital for evaluation and are found to have potassium levels of 5.5 mEq/L and above.

Intervention: Single dose of 5 units of intravenous insulin over 30 minutes with 50 ml of Dextrose 50%.

Clinical Measurement: Mean reduction of potassium level using the main laboratory results at 2 hours from insulin/dextrose administration. Hypoglycemia will be followed by a bedside glucometer.

Outcome: reduction of potassium level at 2 hours from medication administration and medication safety.

ELIGIBILITY:
Inclusion Criteria:

* Hyperkalemia patients with lab potassium levels equal to or more than 5.5 mEq/L (≥ 5.5 mEq/L)+.
* Adult: age 18 years or more.
* Agreed to participate in the study.

  * If an investigator decides to start anti-hyperkalemia medications based on the VBG/ABG patient can be enrolled but if the main laboratory value is less than 5.5 mEq/L patients will be excluded

Exclusion Criteria:

* Cardiac arrest
* Hyperglycemia with random blood sugar 20 mmol/L (13) or with acute diabetic complications like Diabetic Ketoacidosis / Hyperosmolar Hyperglycemic State.
* Hypoglycemia with random blood sugar (RBS) ≤ 3.89 mmol/l in Diabetic patients and less than 3 mmol/l in non-diabetic patients.
* Allergies for any medication in the protocol.
* Pregnancy.
* Hemolyzed potassium level as reported by the main lab.
* Hemolysis, Tumor lysis syndrome, or Rhabdomyolysis due to the ongoing release of potassium.
* Acidosis with a pH less than 7.1 will require Sodium bicarbonate (NaHO3).
* A patient who will need urgent Furosemide (Lasix), and or dialysis during the study period of 2 hours.
* Refused to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
To study the efficacy of two intravenous insulin doses (5 units and 10 units) in reducing serum potassium level in patients receiving hyperkalemia treatment using the main laboratory measurements. (the aim of reduction of 0.6 mmol/l +/- 0.2 mmol/L) (1). | At 2 hours from administration of medications
  Once the baseline potassium identified 5.5 mmol/L or more patient will be enrolled after taken an informed consent. Blood sample will be collected and send to the main laboratory for analysis at two hours from medications administration. The efficacy of the 2 doses of insulin in reducing potassium level will be measured at 2 hours from administration of medications by comparing the amount of changes of potassium level at two hours from baseline level.
  - The main laboratory result will be used to measure and follow the patients. results will be reported in mmol/L.

SECONDARY OUTCOMES:
Study the mean difference of the response to the anti-hyperkalemic measures based on the level of initial potassium (serum potassium before given any medications - At baseline). | 2 hours from administration of medications
  (The investigators will categorize potassium levels into groups mild (5.5-6 mmol/l), moderate (6-6.5 mmol/l), and severe (>6.5 mmol/l) and will see the mean difference in reduction in potassium level between the 2 doses).
Association of mean potassium reduction with initial blood sugar level on potassium reduction | 2 hours from administration of medications
  The investigators will categorize blood sugar into groups: Below 10mmol/L, 10.1-14.9 mmol/L, and 15 - 19.9mmol/L among each group the investigators will see the mean potassium reduction levels.
Incidence of hypoglycemia (random blood sugar (RBS) ≤ 3.89 mmol/l in Diabetic patients and less than 3 mmol/l in non-diabetic patients) (12) and risk factor Characteristics of patients with a higher risk of developing hypoglycemia | 2 hours from administration of medications
  The investigators will investigate which group of patients will have a high risk of hypoglycemia ((e.g.: initial Glucose level, initial creatinin/renal function, comorbidities, type of dialysis….

CONTACTS AND LOCATIONS:
Overall Officials: Suad Al-Abri, Principal Investigator — Sultan Qaboos University hospital
Locations (1):
- Sultan Qaboos University hospital, Seeb, Muḩāfaz̧at Masqaţ, Oman

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Verdier M, DeMott JM, Peksa GD. A comparison of insulin doses for treatment of hyperkalaemia in intensive care unit patients with renal insufficiency. Aust Crit Care. 2022 May;35(3):258-263. doi: 10.1016/j.aucc.2021.05.004. Epub 2021 Jun 21. PMID 34167889
- [Background] Ron M. Walls, MD. Hyperkalemia. Rosen emergency medince Concepts and Clinical practice. 9th. Philadelphia : Elsevier, 2018, 117, pp. 1516 - 1519.
- [Background] Judith E. Tintinalli, MD, MS. Hyperkalemia. Tintinalli's Emergency Medicine a comprehensive study guide. 9th. s.l. : McGraw-Hill Education, 2020, 17, p. 89.
- [Background] McNicholas BA, Pham MH, Carli K, Chen CH, Colobong-Smith N, Anderson AE, Pham H. Treatment of Hyperkalemia With a Low-Dose Insulin Protocol Is Effective and Results in Reduced Hypoglycemia. Kidney Int Rep. 2017 Oct 24;3(2):328-336. doi: 10.1016/j.ekir.2017.10.009. eCollection 2018 Mar. PMID 29725636
- [Background] Moussavi K, Nguyen LT, Hua H, Fitter S. Comparison of IV Insulin Dosing Strategies for Hyperkalemia in the Emergency Department. Crit Care Explor. 2020 Apr 29;2(4):e0092. doi: 10.1097/CCE.0000000000000092. eCollection 2020 Apr. PMID 32426734
- [Background] LaRue HA, Peksa GD, Shah SC. A Comparison of Insulin Doses for the Treatment of Hyperkalemia in Patients with Renal Insufficiency. Pharmacotherapy. 2017 Dec;37(12):1516-1522. doi: 10.1002/phar.2038. Epub 2017 Nov 27. PMID 28976587
- [Background] Moussavi K, Garcia J, Tellez-Corrales E, Fitter S. Reduced alternative insulin dosing in hyperkalemia: A meta-analysis of effects on hypoglycemia and potassium reduction. Pharmacotherapy. 2021 Jul;41(7):598-607. doi: 10.1002/phar.2596. Epub 2021 Jun 1. PMID 33993515
- [Background] Harel Z, Kamel KS. Optimal Dose and Method of Administration of Intravenous Insulin in the Management of Emergency Hyperkalemia: A Systematic Review. PLoS One. 2016 May 5;11(5):e0154963. doi: 10.1371/journal.pone.0154963. eCollection 2016. PMID 27148740
- [Background] Garcia J, Pintens M, Morris A, Takamoto P, Baumgartner L, Tasaka CL. Reduced Versus Conventional Dose Insulin for Hyperkalemia Treatment. J Pharm Pract. 2020 Jun;33(3):262-266. doi: 10.1177/0897190018799220. Epub 2018 Sep 6. PMID 30189765
- See also: David B Mount, MD. Causes and evaluation of hyperkalemia in adults — https://www.uptodate.com/contents/causes-and-evaluation-of-hyperkalemia-in-adults
- See also: Treatment and prevention of hyperkalemia in adults — https://www.uptodate.com/contents/treatment-and-prevention-of-hyperkalemia-in-adults?search=Treatment%20and%20prevention%20of%20hyperkalemia%20in%20adults&source=search_result&selectedTitle=1~150&usage_type=default&display_rank=1
- See also: Hyperkalemia Treatment & Management — https://emedicine.medscape.com/article/240903-treatment
- See also: Hypoglycemia in adults without diabetes mellitus: Clinical manifestations, diagnosis, and causes — https://www.uptodate.com/contents/hypoglycemia-in-adults-without-diabetes-mellitus-clinical-manifestations-diagnosis-and-causes
- See also: Hyper K recognition and treatment of Hyperkalemia in the ED. American College of Emergency Physicians. — https://www.acep.org/patient-care/hyperk/

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/23/NCT06036823/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2023-08-03): https://cdn.clinicaltrials.gov/large-docs/23/NCT06036823/SAP_001.pdf